CLINICAL TRIAL: NCT02130973
Title: The Treatment of Osteoporosis Using a Combination of Teriparatide (Forteo) and Denosumab
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Health Research, Inc. (Other)
Responsible Party: Principal Investigator, Felicia Cosman, M.D., Professor of Clinical Medicine, Health Research, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMG 10-05
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Osteoporosis
Keywords: teriparatide; Forteo; Denosumab; Prolia; bone density; treatment
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Clinical Practice Regimen (Active Comparator): Standard Clinical Practice (Daily) Regimen: 18 months of daily subcutaneous Forteo followed by denosumab therapy for 18 months (18 months of Forteo then 3 injections of Prolia at 18, 24 and 30 months).
  Interventions: Drug: Standard Clinical Practice Regimen
- Experimental (cyclic) regimen (Experimental): Experimental (Cyclic) Regimen: three separate 6-month cycles of daily subcutaneous Forteo, each followed by one subcutaneous injection of Prolia (Forteo from 0 to 6 months, and then from 12 to 18 months and then from 24 to 30 months, for a total dose of 18 months; 3 injections of Prolia at 6, 18 and 30 months).
  Interventions: Drug: Experimental Cyclic Regimen

INTERVENTIONS:
Drug: Standard Clinical Practice Regimen — Standard Clinical Practice Regimen
  Other Names: 18 months Forteo followed by 18 months Prolia
  Arms: Standard Clinical Practice Regimen
Drug: Experimental Cyclic Regimen — Experimental Cyclic Regimen
  Other Names: three separate 6 month cycles of daily Forteo, each followed by one of Prolia
  Arms: Experimental (cyclic) regimen

SUMMARY:
This is a three-year study to evaluate the effect of sequential therapy of Forteo (teriparatide) and denosumab on bone density at the spine, hip, leg and forearm.

DETAILED DESCRIPTION:
In order to maximize the early anabolic effect with teriparatide (TPTD), and to avoid the development of tachyphylaxis to the continued daily administration of TPTD beyond 6 months, cyclic therapy might be optimal. Since Denosumab (Prolia) is a potent antiresorptive agent with a rapid off-effect, it might be the optimal agent to help maximize bone gains with cyclic TPTD/antiresorptive therapy. Our primary hypothesis is that the increment in bone density of the spine by DXA will be greater in women randomized to receive the cyclic sequential regimen (three separate 6 month cycles of daily subcutaneous TPTD, each followed by one subcutaneous injection of Denosumab) compared with daily sequential therapy (18 months of daily subcutaneous TPTD followed by Denosumab therapy for 18 months).

ELIGIBILITY:
Inclusion Criteria:Subjects should be postmenopausal >age 45, and of any racial origin. They must not be on any osteoporosis medication. They should be willing to participate for the duration of the study and have no physical or psychological illness that would prohibit them from participating. Pregnant women, protected individuals (institutionalized), and those unable to give informed consent will not be recruited. Exclusion criteria are detailed below.

Subjects who meet initial pre-screening criteria will present for an on site screening visit and have a full medical history, brief physical exam, BMD and lab evaluation to confirm eligibility. Osteoporosis will be defined by DXA BMD T-Score < -2.5 at lumbar spine (at least 2 evaluable vertebrae between L1 and L4), or total hip or femoral neck. In addition, women with confirmed vertebral deformity on radiograph or lateral DXA image, or prior osteoporosis-related fracture at age >45 along with a DXA BMD T-Score < -1.5 at one or more skeletal sites will be eligible to participate.

Exclusion Criteria:

* The use of drugs known to affect skeletal or calcium homeostasis.
* Multiple vertebral fractures or severe lumbar degenerative changes with fewer than 2 evaluable lumbar vertebrae
* Current use of anti-resorptive medicines

  * Use of Hormone/Estrogen Therapy, raloxifene or calcitonin within the past 3 months
  * Use of oral bisphosphonate for more than 4 months within the past 2 years or more than 5 years total cumulative bisphosphonate use in the past 10 years
  * Use of intravenous ibandronate within the past 18 months
  * Use of intravenous zoledronic acid within the past 4 years
  * A history of a symptomatic renal stone within the past 3 years or history of multiple symptomatic renal stones
  * Skeletal Disorders other than osteoporosis including: Hypercalcemia, hyperparathyroidism, Paget's Disease or osteomalacia
  * Untreated or uncontrolled thyroid disease
  * Elevated Bone Specific Alkaline Phosphatase level
  * History of external or internal radiation therapy
  * Renal insufficiency with estimated GFR below 30 ml/min
  * Liver function tests (ALT/AST) more than 1.5 times the upper limit of normal
  * Clinically significant hyperuricemia or active gout
  * Any contraindications to receipt of Teriparatide or Denosumab (including hypocalcemia)
  * History of an atypical fracture of the femoral shaft

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
spine bone density | 3 years

SECONDARY OUTCOMES:
bone mineral density of the hip, wrist, total body and lateral spine and CT of arm and leg | 3 years
  Bone mineral density testing of multiple skeletal sites and peripheral QCT with high resolution of the leg and arm

OTHER OUTCOMES:
bone turnover | 3 years
  Measurement of bone formation and bone resorption

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Cosman, M.D., Principal Investigator — Helen Hayes Hospital
Locations (1):
- Helen Hayes Hospital, West Haverstraw, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cosman F, McMahon D, Dempster D, Nieves JW. Standard Versus Cyclic Teriparatide and Denosumab Treatment for Osteoporosis: A Randomized Trial. J Bone Miner Res. 2020 Feb;35(2):219-225. doi: 10.1002/jbmr.3850. Epub 2019 Oct 23. PMID 31419313